CLINICAL TRIAL: NCT00594724
Title: Improving Therapeutic Outcomes in the Tongue Carcinoma Patient: Assessment of Adaptation Using Functional Magnetic Resonance Imaging and Diffusion Tensor Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rockefeller University (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-093
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Tongue Carcinoma
Keywords: Tongue; Carcinoma; Cancer; 02-093
MeSH Terms: conditions — Tongue Neoplasms; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Adaptation Using Functional Magnetic Resonance Imaging and Diffusion Tensor Imaging

SUMMARY:
The purpose of this study is to see how the brain re-learns to control the tongue in speaking and swallowing when either portions of the tongue have been removed, or when the tongue has been treated with radiation, in order to treat cancer. We hope the results of this study will help us to improve healing for patients who are being treated for cancer of the tongue.

When patients with cancer of the tongue are treated by removing parts of the tongue (surgery) or by destroying the cancer with radiation to the tongue, they have significant difficulty speaking and swallowing after such treatments. At this time, patients who have been treated for cancer of the tongue re-learn speaking and swallowing through exercises taught by a speech pathologist.

What is needed is information on how the brain re-learns to control speaking and swallowing so that we can help these patients re-learn faster after their treatments.

DETAILED DESCRIPTION:
The purpose of this investigation is to determine cortical mechanisms of adaptation to surgical or radiation treatment to the tongue. This study will use a non-invasive imaging technique, Functional Magnetic Resonance Imaging (fMRI), to investigate cortical responses to partial glossectomy or radiation therapy for treatment of a tongue malignancy. Patients with Stage I-IV (AJCC) malignancies of the tongue who are treated with surgery and or radiation therapy will be imaged using fMRI pre-operatively and at approximately six months postoperatively.

Patterns of brain activity from the fMRI studies will be compared with matched healthy control subjects. The results of this investigation will provide needed information on both central and peripheral mechanisms of adaptation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the tongue carcinoma patients:

* Primary malignancy of the oral or base of tongue, Stage I-IV of AJCC staging system, planned for surgical or radiation therapy.

Inclusion criteria for the healthy subjects:

* Healthy adult subjects between the ages of 21-75 years.

Exclusion Criteria:

Exclusion criteria for the tongue carcinoma patients include the following:

* History of significant psychiatric condition (e.g. schizophrenia, obsessive-compulsive disorder, significant dementia),
* History of the following neurological conditions: CVA, seizure disorders, demyelinating conditions, systemic neuromuscular disorders, cerebral palsy, Alzheimer's disease.
* History of previous moderate to severe traumatic brain injury.
* History of significant cardiovascular, respiratory, gastrointestinal or renal disease (e.g.myocardial infarction within the previous 12 months, significant vaso-occlusive disease,severe or advanced asthma, COPD, emphysema, gastroesophageal reflux disease, or renal compromise)
* History of achalasia
* History of other neoplasms involving the brain, head and neck, or gastrointestinal system.
* History of dysphagia, odynophagia, or aphasia unrelated to present illness.
* History of significant claustrophobic reactions.
* Standard contraindications to MR examinations (e.g. implanted stimulators).

Exclusion criteria for the healthy subjects includes the all of the conditions listed for the tongue:

* Carcinoma patients and additionally includes history of significant surgery or previous radiation therapy to the head and neck
* Previous history of dysphagia, odynophagia, aphasia, pregnancy,and standard contraindications to MR examinations.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2002-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To utilize fMRI to characterize adaptation to alterations in tongue morphology & function following either surgical therapy, or radiation/chemotherapy to tongue in patients undergoing treatment of malignancies involving the tongue. | 7 years

SECONDARY OUTCOMES:
Determine relationship between mechanisms of adaptation at level of central nervous system to alterations in function in the tongue. | 7 years
Determine changes in cortical activity in representation of tongue movement that occur pre and post-treatment. | 7 years
Determine the central neural response to direct peripheral rehabilitation strategies. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Peck, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org